CLINICAL TRIAL: NCT01700790
Title: A Pharmacokinetic Study of Super-boosted Lopinavir/Ritonavir in Combination With Rifampin in HIV-1-infected Patients With Tuberculosis.
Brief Title: Pharmacokinetic Study of Super-boosted Lopinavir/Ritonavir Given With Rifampin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No Further Funding
Sponsor: University of Miami (Other)
Collaborators: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Catherine Boulanger, Associate of Professor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100325
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2018-12

CONDITIONS: AIDS; Tuberculosis
Keywords: HIV; AIDS; Tuberculosis; Rifampin; Lopinavir; Pharmacokinetic
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — lopinavir-ritonavir drug combination; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lopinavir/ritonavir and ritonavir (Experimental): Two tablets of twice daily of Lopinavir/ritonavir 200 mg/50mg with 3 tablets of ritonavir 100 mg of twice daily given with rifampin 600 mg daily.
  Interventions: Drug: Lopinavir/ritonavir and ritonavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir and ritonavir — Two tablets twice daily of Lopinavir/ritonavir 200 mg/50mg with 3 capsules of ritonavir 100 mg twice daily given with rifampin 600 mg daily
  Other Names: Kaletra; Norvir

SUMMARY:
The object of this study is to evaluate the pharmacokinetic interactions, short term safety and efficacy of standard dose lopinavir/ritonavir 200mg/50 (two tablets twice daily) given with ritonavir 100 mg three tablets twice daily given in combination with rifampin in HIV-infected persons with tuberculosis

DETAILED DESCRIPTION:
This will be an open label non-randomized pharmacokinetic study of 10-12 HIV-infected patients co-infected with Mycobacterium tuberculosis.

Enrollment: Potential subjects with active tuberculosis who have tolerated a rifampin containing regimen for at least 2 weeks. Potential subjects will be referred from the surrounding communities to Laboratorio de Pesquisa Clinica em Micobacterioses(LAPCLINTB)

Visit 1: Subjects will then be started on lopinavir/ritonavir containing HAART regimen with standard twice daily dosing. Ritonavir 100 mg capsules will be added to the regimen and the dose escalated until the patient is taking 3 capsules twice daily. The time between enrollment and visit 1 will be determined by the treating physician.

Visit 2: They will return about 1 week after dose escalation has been completed to sample lopinavir and rifampin concentrations.

Visit 3: Subject will return in 2 weeks to have repeat to review results of lopinavir concentrations and response to therapy. Ritonavir will be adjusted as needed.

Visit 4: Subject will then return in 4 weeks for last visit for evaluation. Lopinavir and rifampin PK will be done.

ELIGIBILITY:
* Antiretroviral naive
* If not antiretroviral naïve they must meet the following criteria:

  * Taking Kaletra containing regimen with suppressed viral load.
  * Taking an NNRTI or integrase containing regimen without prior history of use of PI for more than 2 weeks
  * Taking an NNRTI or integrase containing regimen with prior exposure to PI greater than 2 weeks. It must be clearly stated in the source document that PI was switched to another agent for convenience.
  * Taking another PI containing regimens with suppressed viral load. It must be clearly stated in source document that if another PI was used for greater than 2 weeks the regimen was switched to another agent for convenience. Subjects with prior history of PI use may be enrolled, if there is a genotype showing no resistance to Kaletra Other Inclusion criteria
* Be at least 18 years of age and able to give informed consent.
* Diagnosed with TB by criteria per Brazilian Ministry of Health
* Have a good clinical response to TB.
* Tolerating tuberculosis therapy containing rifampin for the 2 weeks prior to screening,except for persons taking protease inhibitors at time of diagnosis of TB.,. Subjects taking protease inhibitors will be screened and initiate visit 1 within 3 days of starting TB medication
* HIV positive with documentation present in source document.
* Have a CD4 cell count greater than 50 cells/mm3if not taking ART. Persons with cd4 < 50 may be enrolled, if it is felt that in the best interest of the patient, that enrollment in the study will allow for quicker initiation of antiretroviral therapy than referral to another treatment center.

Exclusion Criteria:

* Non-compliance with DOTPlus. Alternatively DOT can be done by telephoning patient on a daily basis 5 times a week and having patient annotate taking drug in a log which would be reviewed by clinic staff
* History of being treated for tuberculosis in the prior 2 years unless there is DST, including PCR testing, showing sensitivity to rifamycin.
* Known hypersensitivity to rifampin or rifabutin.
* Liver enzymes greater than 2 times ULN.
* Bilirubin greater than 2 times ULN.
* Serum creatinine greater than 3 times ULN.
* Hemoglobin less than 7.0 gms even if receiving erythropoietin.
* Absolute neutrophil count less than 750 cells/mm3 even if receiving G-CSF.
* Fasting triglycerides greater than 400 mg/dL.
* Fasting cholesterol > 1.6 upper limits of normal.
* GI intolerance of tuberculosis medications requiring discontinuation of tuberculosis medications.
* Fasting glucose greater 150 mg/dL.
* Pregnant women.
* Use of one of the prohibited medications
* Any condition that the investigators feel could compromise the use of the current medication.
* Have a CD4 cell count of 50 cells/mm3or less
* Hepatitis B or C infection
* Alcohol or illicit drug use, which in the investigators opinion may affect participation in study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with expected pre dose concentration of lopinavir. | Weeks 2 and 8: lopinavir time points at hours 0, 2, 4, 6 and 8.
  The expected pre dose concentration of lopinavir is >1.0 mcg/mL.

SECONDARY OUTCOMES:
Proportion of patients with successful treatment of HIV therapy. | Approximately 10-12 weeks
  HIV failure will be defined as failure to drop the viral load by 0.5 log 10 copies/mL drop by week 4 of treatment and a viral load drop >1 log 10 copies/ml by week 8.
Proportion of patients with expected AUC of rifampin | Approximatley 10-12 weeks
  The expected AUC of rifampin is 44-70 mcg•h/mL
Proportion of patient with success of tuberculosis therapy | Approximatly 10-12 weeks
  Success of treatment using criteria established by the Brazilian National Ttuberculosis Program.
Proportion of patients with expected Cmax and AUC of lopinavir | 10-12 weeks
  The expected Cmax of lopinavir is 6-14 mcg/mL. The expected AUC lopinavir is 56-130 µg•h/mL
Proportion of patients with expected Cmax of rifampin. | Weeks 2 and 8: rifampin time points at hours 0, 2, 4, 6 and 8.
  Expected maximum concentration of rifampin is 8-24 mcg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Boulanger, MD., Principal Investigator — University of Miami Miller Medical School of Medicine; Valeria Calvicanti Rolla, MD, Principal Investigator — Oswaldo Cruz Foundation
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas - Fiocruz(INI), Laboratorio de Pesquisa Clinica em Micobacterioses(LAPCLINTB), Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ren Y, Nuttall JJ, Egbers C, Eley BS, Meyers TM, Smith PJ, Maartens G, McIlleron HM. Effect of rifampicin on lopinavir pharmacokinetics in HIV-infected children with tuberculosis. J Acquir Immune Defic Syndr. 2008 Apr 15;47(5):566-9. doi: 10.1097/QAI.0b013e3181642257. PMID 18197120
- [Background] la Porte CJ, Colbers EP, Bertz R, Voncken DS, Wikstrom K, Boeree MJ, Koopmans PP, Hekster YA, Burger DM. Pharmacokinetics of adjusted-dose lopinavir-ritonavir combined with rifampin in healthy volunteers. Antimicrob Agents Chemother. 2004 May;48(5):1553-60. doi: 10.1128/AAC.48.5.1553-1560.2004. PMID 15105105
- [Derived] Boulanger C, Rolla V, Al-Shaer MH, Peloquin C. Evaluation of super-boosted lopinavir/ritonavir in combination with rifampicin in HIV-1-infected patients with tuberculosis. Int J Antimicrob Agents. 2020 Feb;55(2):105840. doi: 10.1016/j.ijantimicag.2019.10.021. Epub 2019 Nov 5. PMID 31704214